CLINICAL TRIAL: NCT07039058
Title: Brief Dialectical Behavior Therapy-Skills Training for Coping With Suicidal Ideation: A Randomized Controlled Trial
Brief Title: Brief DBT Skills Training for Coping With Suicidal Ideation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not initiated due to lack of resources.
Sponsor: Muhammed Ali Boztepe (Other)
Responsible Party: Sponsor-Investigator, Muhammed Ali Boztepe, Clinical Psychology Master's Student, Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BriefDBT-ST30/05/2025
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Suicide Ideation; Coping Skills; Emotion Regulation
Keywords: Dialectical Behavior Therapy; Skills Training; Suicide ideation; Randomized
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Dialectical Behavior Therapy-Skills Training (Experimental)
  Interventions: Behavioral: Brief Dialectical Behavior Therapy-Skills Training
- Relaxation control group (Active Comparator)
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Behavioral: Brief Dialectical Behavior Therapy-Skills Training — The intervention is administered in a single session, lasting approximately 60 minutes and conducted in person. It is important to note that there are no ongoing sessions.
  In the intervention, participants are provided with 5 basic skills of Dialectical Behavior Therapy: 1) mindfulness, 2) mindfulness of current emotions, 3) opposite-to-emotion action, 4) distraction, and 5) changing body chemistry. These strategies are grouped under 3 categories: 1) Mindfulness, 2) Emotion regulation (mindfulness of current emotions, opposite-to-emotion action), 3) Tolerating distress (distraction, changing body chemistry). These skills are not designed to treat or solve the crisis. The main aim is to provide effective coping mechanisms that can be implemented quickly before the crisis escelates, to help overcome the intense emotional pain and keep the person alive.
  Arms: Brief Dialectical Behavior Therapy-Skills Training
Behavioral: Relaxation — The control group will be subjected to a relaxation exercise, with the objective of managing participant expectations, researcher attention/interest, and time spent, as well as providing a coping strategy for stress.
  Arms: Relaxation control group

SUMMARY:
The goal of this clinical trial is to learn if Brief Dialectical Behavior Therapy Skills Training (DBT-BST) can prevent suicidality in adults. The main questions it aims to answer are:

* Does DBT-BST provide coping strategies (e.g., emotion regulation) to participants with suicidal ideation?
* Does DBT-BST lower participants' suicide ideation?

Researchers will compare DBT-BST to relaxation to see if DBT-BST works to reduce suicidal ideation.

Participants will:

* Receive DBT-BST in a single 60-minute, in-person, individual session.
* Be asked to use these skills as self-help and for crisis prevention.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years of age or older
* having suicidal ideation in the last 3 months
* not having received any psychological treatment in the last 1 month
* living in Aydın/Türkiye where the intervention will be implemented
* giving consent for participation

Exclusion Criteria:

* not speaking Turkish
* loss or trauma in the last 1 year
* pharmacological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Suicidality at 1 Month as Assessed by Suicide Probability Scale | From enrollment to the end of intervention at 1 week and follow-up at 1 month
  36 is equivalent to the lowest suicidality, and 144 indicates the highest suicidality.
Change from Baseline in the Suicidal Cognitions at 1 Month as Assessed by Suicide Cognitions Scale | From enrollment to the end of intervention at 1 week and follow-up at 1 month
  18 is equivalent to the lowest suicidal cognitions, and 90 indicates the highest suicidal cognitions.
Change from Baseline in the Hopelessness at 1 Month as Assessed by Beck Hopelessness Scale | From enrollment to the end of intervention at 1 week and follow-up at 1 month
  Zero is equivalent to the lowest hopelessness, and 20 indicates the highest hopelessness.
Change from Baseline in the Emotion Regulation Skills at 1 Month as Assessed by Emotion Regulation Skills Questionnaire | From enrollment to the end of intervention at 1 week and follow-up at 1 month
  Zero is equivalent to the lowest emotion regulation skills, and 108 indicates the highest skills.
Change from Baseline in the Difficulties in Emotion Regulation at 1 Month as Assessed by Difficulties in Emotion Regulation Scale-16 | From enrollment to the end of intervention at 1 week and follow-up at 1 month
  16 is equivalent to the lowest difficulties, and 80 indicates the highest difficulties in emotion regulation.

SECONDARY OUTCOMES:
Change from Baseline in the Depression, Anxiety, and Stress at 1 Month as Assessed by Depression Anxiety Stress Scale-21 (DASS-21) | From enrollment to the end of intervention at 1 week and follow-up at 1 month
  Higher points are equivalent to higher symptoms as assessed by the related subscale of DASS-21. Each subscale ranges from 0 to 28.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Suicide and Stress Research Laboratory, Aydin, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided